CLINICAL TRIAL: NCT02577302
Title: Multi-center, Prospective, Randomized, Controlled, Non-Inferiority, Clinical Trial of Chronic Afferent Nerve Stimulation (CAN-Stim) of the Tibial Nerve Versus Sacral Nerve Stimulation (SNS) in the Treatment of Urinary Urgency Incontinence Resulting From Refractory Overactive Bladder (OAB)
Brief Title: CAN-Stim Compared to SNS in Treatment of Urinary Urgency Incontinence With Wireless Neuromodulation Technology
Acronym: PROTECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uro Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30-00137
Record Dates: First submitted 2015-10-12; First posted 2015-10-16 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Urinary Incontinence, Urge
Keywords: Chronic Tibial nerve stimulation; Wireless PNS; neuromodulation
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Controlled, Non-Inferiority
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- CAN-Stim Group - CAN-Stim System (Experimental): Intervention: tibial medical device
  Subjects randomized to this group will have the Protect CAN-Stim System tibial medical device implanted for the duration of the study.
  Interventions: Device: CAN-Stim - Protect CAN-Stim System
- SNS Group - Interstim® System (Active Comparator): Intervention: SNS Medical device
  Subjects randomized to SNS will have their Stage I device implanted and tested during a 2-week period. Stage I will have a tined, quadripolar lead placed in the S3 (preferred) or S4 (alternate) foramen in the standard fashion using fluoroscopic guidance and motor response. Motor responses can include a contraction of the levators ("bellows" response) with or without plantar flexion of the great toe. Subjects who are not demonstrating an appropriate motor response will not have the device implanted and will be exited from the study.
  Interventions: Device: SNS - InterStim® System

INTERVENTIONS:
Device: CAN-Stim - Protect CAN-Stim System — CAN-Stim subjects will be implanted unilaterally (implantation side is up to the investigators discretion) with the CAN-Stim System. Subjects will be educated on the use of the transmitter and programmer. Therapy will be delivered for a minimum of 8 hours per day for 2 weeks. Subjects who are considered a responder at the 2-week follow-up, will continue therapy and followed for a total of 12 months.
  Arms: CAN-Stim Group - CAN-Stim System
Device: SNS - InterStim® System — Subjects randomized to SNS will have their Stage I device implanted and tested during a 2-week period. Stage I will have a tined, quadripolar lead placed in the S3 (preferred) or S4 (alternate) foramen in the standard fashion using fluoroscopic guidance and motor response. Motor responses can include a contraction of the levators ("bellows" response) with or without plantar flexion of the great toe. Subjects who are not demonstrating an appropriate motor response will not have the device implanted and will be exited from the study.Therapy will be delivered for a minimum of 8 hours per day for 2 weeks. Subjects who are considered a responder at the 2-week follow-up, will receive a full implant and followed for a total of 12 months.
  Arms: SNS Group - Interstim® System

SUMMARY:
This is a prospective, randomized, controlled, multi-center, study in which 150 evaluable subjects will be randomized 1:1 to receive either a Protect CAN-Stim or SNS InterStim® system. Subjects from both groups will immediately start with therapy. The primary endpoint is a ≥ 50% reduction in number of incontinence episodes associated with urgency at the 3-month visit, with additional measurements assessed at 14 days, 1, 6, 9 and 12-months.

DETAILED DESCRIPTION:
Subjects will be randomized at baseline to either CAN-Stim or SNS InterStim® after inclusion and exclusion criteria have been met, 150 subjects will be randomized in to either arm of the study (89 subjects each arm).

At the following visit, CAN-Stim subjects will be immediately implanted unilaterally with a permanent device (implantation side up to investigators discretion). During implantation, the subject should feel pulsation in their foot with or without toe flexion, confirming stimulation of the tibial nerve. Subjects not achieving this motor response will not have the device implanted and will be exited from the study. Implanted subjects will be educated on the use of the transmitter and programmer. Programming parameters will be set and therapy will be delivered for a minimum of 8 hours per day for 2 weeks. Programming changes can be done as needed during this time period to maximize clinical response. At the 2-week visit, diaries will be reviewed and confirmed for accuracy and discrepancies and the number of urgency incontinence episodes will be calculated and compared to baseline diaries. Subjects who are considered a responder at the 2-week follow-up visit (>50% improvement in urgency related incontinence episodes) will continue therapy and followed for a total of 12 months with primary outcomes assessed at 3 months. Non-responders will be offered an explant of the device and will exit the study. Subjects having less than 50% improvement may choose to keep the device. These subjects will be followed for adverse events with phone calls at 3, 6 and 12 months.

Subjects randomized to SNS will have their Stage I device implanted and tested during a 2-week period. Stage I will have a tined, quadripolar lead placed in the S3 (preferred) or S4 (alternate) foramen in the standard fashion using fluoroscopic guidance and motor response. Motor responses can include a contraction of the levators ("bellows" response) with or without plantar flexion of the great toe. Subjects who are not demonstrating an appropriate motor response will not have the device implanted and will be exited from the study. Subjects, who respond intraoperatively, will have the extension lead connected and externalized in the standard fashion. Subjects may have their InterStim® activated 24 hours/day, but a minimum of 8 hours per day for 2 weeks is required to remain in the study. Programming changes can be done as needed during this time period to maximize the clinical effect. At the 2-week visit, diaries will be reviewed and confirmed for accuracy and clarified for discrepancies and the number of urgency incontinence episodes will be calculated and compared to baseline diaries. Patients achieving a clinical response (>50% improvement in urgency related incontinence episodes) will undergo implantation of a pulse generator and removal of the percutaneous extension lead. The IPG will be programmed in the standard fashion using settings that were working for the patient during the 2-week trial. Subjects implanted with the InterStim® device will be monitored for a total of 12 months with primary outcomes assessed at 3 months. Non-responders will be offered an explant of the device and will exit the study. Subjects having less than 50% improvement may choose to keep the device. These subjects will be followed for adverse events with phone calls at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of overactive bladder with urgency urinary incontinence or mixed incontinence (urge and stress) with predominate urge, as confirmed by the MESA questionnaire;
* Women and men ≥ 18 years of age;
* Women of child-bearing age willing to practice birth control;
* At least 4 incontinent episodes associated with urgency on a 3-day voiding diary;
* At least 10 voids per day;
* Average urgency score of at least 2 as measured with IUSS on a 3-day voiding diary;
* Self-reported bladder symptoms present > 6 months;
* Documented failure of an adequate trial of first and second line therapy;
* Off all antimuscarinics and beta-3 adrenergic agonists for at least 2 weeks prior to enrollment;
* If on Tricyclic antidepressants, dosage must be stabilized for at least 3 months;
* Have no active urethral obstruction/stricture, bladder calculi or bladder tumor based on medical history;
* Normal upper urinary tract function based on medical history;
* Based on the medical opinion of the Investigator, there is no evidence of anatomic abnormalities that could jeopardize the placement of the device or pose a hazard to the subject;
* Based on the medical opinion of the Investigator, subject is willing and able to operate the patient programmer, recharging equipment, diary and has the ability to undergo study assessments and provide accurate responses;
* Based on the medical opinion of the Investigator, subject is a good surgical subject for the implant procedure;
* Capable of giving informed consent;
* Capable and willing to follow all study related procedures.

Exclusion Criteria:

* An active implantable electronic device regardless of whether stimulation is ON or OFF;
* Pregnant as confirmed by a urine pregnancy test or plan to become pregnant during the following 12 months period;
* Primary complaint of stress urinary incontinence;
* Less than 1 year post-partum and/or are breast-feeding;
* Neurogenic bladder (i.e. Multiple sclerosis, Parkinson's, Spinal Cord Injury);
* Patients with spinal hardware that would limit access to the sacrum;
* Botox use in bladder or pelvic floor muscles in the past nine months;
* Have a post-void residual urine volume >150 cc at baseline;
* Current urinary tract infection (UTI);
* Previous treatment with sacral neuromodulation;
* Previous treatment with percutaneous tibial nerve stimulation, pelvic floor muscle stimulation, or biofeedback within the past 60 days;
* Conditions requiring Magnetic Resonance Imaging (MRI) evaluation or diathermy procedures;
* Inability to operate the CAN-Stim System or InterStim System;
* Diabetes with peripheral nerve compromise or severe uncontrolled diabetes (HbA1C 8.5 or greater);
* History of coagulopathy or bleeding disorder;
* History of pelvic pain as primary diagnosis (VAS score of > 4) at baseline;
* Anatomical restrictions such that device placement is not possible;
* Are currently participating or have participated within the past 30 days in any clinical investigation involving or impacting urinary or renal function;
* Have a life expectancy of less than 1 year;
* Cannot independently comprehend and complete the questionnaires and diaries;
* Deemed unsuitable for enrollment by the investigator based on history or physical examination (including bleeding disorders or anticoagulant medications, and peripheral neuropathy);
* Dependent on wearable, transcutaneous, or other therapeutic medical device (examples: glucose monitor, TENS) for treatment of a disease or disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Response rate: a ≥ 50% reduction in number of urgency related incontinence episodes | 3 Months
  The primary efficacy endpoint is defined as a ≥ 50% reduction in number of urgency related incontinence episodes at 3 months post-implant of the CAN-Stim system compared to SNS InterStim® system therapy. The number of urgency incontinent episodes per day is taken as an average of two 3-day consecutive bladder diaries, with at least 24 hours between when the first diary ends and the second diary begins
device- and procedure-related Adverse Events (AE) | 3 Months
  The safety endpoint is the device- and procedure-related Adverse Events (AE) rate at 3 months in the CAN-Stim and SNS groups.

SECONDARY OUTCOMES:
Response rate: a ≥ 50% reduction in number of urgency related incontinence episodes | 6,12 Months
  The endpoint is defined as a ≥ 50% reduction in number of urgency related incontinence episodes at 6 and 12 months post-implant of the CAN-Stim system compared to SNS InterStim® system therapy. The number of urgency incontinent episodes per day is collected with a voiding diary.
device- and procedure-related Adverse Events (AE) | 6,12 Months
  The safety endpoint is the device- and procedure-related Adverse Events (AE) rate at 6 and 12 months in the CAN-Stim and SNS groups.
Voiding Frequency | 3, 6,12 Months
  The achievement in each subject of a ≥ 50% reduction in the number of voids or a return to normal voiding frequency (< 8 voids/day) from baseline to 3-, 6-, and 12-month follow-up in the CAN-stim group compared to the InterStim® group;
Reduction in degree of urgency | 3, 6,12 Months
  A reduction in the degree of urgency as measured with the Indevus Urgency Severity Scale (IUSS) in the CAN-Stim group compared to the InterStim® group.

OTHER OUTCOMES:
Quality of Life: I-QOL: Quality of Life Scale (I-QOL) | 3, 6,12 Months
  Change in the Urinary Incontinence Quality of Life Scale (I-QOL) in the CAN-Stim group compared to the InterStim® group
Proportion of subjects dry | 3, 6,12 Months
  B. The proportion of subjects dry as measured by the number of incontinence episodes per day associated with urgency as captured on the voiding diary.
Episodes | 3, 6,12 Months
  The number of episodes associated with urgency as illustrated by voiding diaries
Improvement | 3, 6,12 Months
  Global Response Assessment (GRA) will be used to compare the proportion of subjects reporting "moderately" or "markedly improved" responses on all subject visits
OAB | 3, 6,12 Months
  Overactive Bladder Questionnaire Short Form (OAB-Q)
AE's | 6, 12 months
  Adverse events both related or unrelated in the CAN-Stim group compared to the InterStim® group throughout the study

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Tilda Research Inc, Laguna Hills, California
  - Kaiser Permanente, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - Westview Clinical Research, Placentia, California
  - Advanced Urology Institute, Daytona Beach, Florida
  - Baptist Health Miami Cancer Institute, Miami, Florida
  - Florida Urology Partners, Tampa, Florida
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Louis Pain Consultants, St Louis, Missouri
  - Adult & Pediatric Urology, P.C., Omaha, Nebraska
  - Urology - Iris Cantor Men's Health Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Integrated Pain Specialists, Columbus, Ohio
  - University of Oklahoma health Sciences Center, Oklahoma City, Oklahoma
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
upon study completion